CLINICAL TRIAL: NCT05470309
Title: Using a Community-based Participatory Approach to Reduce Disparities in Cervical Cancer Prevention, Screening, and Diagnosis Among Hispanic Women in Cleveland
Brief Title: Community Outreach-based Study to Increase Cervical Cancer Screening Among Hispanic Women in Cleveland
Status: Withdrawn | Type: Observational
Why Stopped: Personnel departure.
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000024
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer Screening; Home HPV Self-Test; In-office Pap Test; Hispanic Women; Cleveland
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study offers Hispanic women who are eligible for cervical cancer screening residing in the Cleveland metropolitan area one of two possible community outreach-based cervical cancer screening modalities, self-collection home HPV test or clinic-based pap test, which is the current standard of care, to assess if these strategies improve cervical cancer screening rates in this population group.

DETAILED DESCRIPTION:
This study is an observational community outreach-based feasibility study. The study intervention that is being evaluated includes two different strategies of cervical cancer screening: 1) a self-collection home HPV test and 2) an in-office pap test. Study subjects who choose the self-collection home HPV test will be provided with the following materials: 1) research information sheet that explains the study objective, the expected timeline of the results, 2) a letter recommending a routine pap test regardless of whether they chose to complete the self-sampling HPV test, 3) educational materials on how to self-collect and return a sample, and 4) a FDA-approved self-sampling kit. Self-collected samples will be tested by the FDA-approved procedure. Study subjects will be asked to choose the screening method of their preference: a self-collection HPV testing kit at home and return the kit within 1 month to the study team or a pap test at a local clinic, which is scheduled within a month. The at-home test only includes vaginal swab and not collection from the cervix. The study team will be notified of the results of HPV test or of pap test and inform the study subjects. If the study subject reports the study team of the loss of her home HPV test kit, it will be recorded as a study outcome of "loss of home HPV test kit". Study subjects who do not return their HPV test kit within 4 weeks will receive 3 reminder calls within a week.

Study subjects who choose an in-office pap test will be scheduled for an annual gynecological exam that includes a pap test at a local clinic that the participant prefers by the study team. The standard-of-care in gynecology at the local clinic involves annual gynecological exam. Study subjects who choose an in-office pap test will receive two appointment reminder calls by the study team a week and three days prior to the scheduled appointment, respectively. No returning of the self-sampling home HPV kit and no show to the scheduled appointment for pap test will be recorded as study outcomes, and these study subjects will be considered enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women aged 30 and 65 years
* Residing in the City of Cleveland

Exclusion Criteria:

* Women who are pregnant
* Had a hysterectomy
* Women who had pap test in the past three years or hrHPV test in the past five years or co-testing (hrHPV + pap test) in the past five years.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Hispanic women aged 30 and 65 years residing in the City of Cleveland who are not pregnant; did not have a hysterectomy; and are due for guideline-recommended cervical cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Receipt of Cervical Cancer Screening | 3 months
  Either return of a mailed home HPV test kit or receipt of in-office Pap test

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Y Eom, PhD, Principal Investigator — MetroHealth Population Health Research Institute
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No